CLINICAL TRIAL: NCT00840645
Title: Long-term Study of YM178: Long Term Study of YM178 in Subjects With Overactive Bladder
Brief Title: A Long-term Study of YM178 in Symptomatic Overactive Bladder Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 178-CL-051
Record Dates: First submitted 2009-02-08; First posted 2009-02-10 (Estimated); Last update posted 2016-01-05 (Estimated); Status verified 2016-01

CONDITIONS: Urinary Bladder, Overactive
Keywords: YM178; Urinary Bladder, Overactive; Mirabegron
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — mirabegron

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1. YM178 (Experimental)
  Interventions: Drug: YM178

INTERVENTIONS:
Drug: YM178 — Oral
  Other Names: Mirabegron

SUMMARY:
The study is intended to test the safety, tolerability, and efficacy of long-term treatment with YM178 in patients with overactive bladder symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Subject has symptoms of overactive bladder for >= 24 wks
* Subject experiences frequency of micturition at average >= 8 times per 24 hrs confirmed by the 3-day patient diary

Exclusion Criteria:

* Subject is breastfeeding, pregnant, or intends to become pregnant during the study
* Subject obviously has stress incontinence
* Subject has an indwelling catheter or practices intermittent self catheterization
* Subject has evidence of symptomatic urinary tract infection, interstitial cystitis, bladder stone, etc
* Subject has an average total daily urine volume > 3000 mL confirmed by patient diary
* Subject has uncontrollable hypertension (SBP >= 180 mmHg or DBP >= 110 mmHg)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2008-12; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Vital signs, AEs, lab tests, ECG, post-void residual volume | 52 weeks

SECONDARY OUTCOMES:
Changes from baseline in the mean number of micturitions/24hrs | 52 weeks
Changes from baseline in the mean number of urinary urgencies/24 hrs | 52 weeks
Changes from baseline in the mean number of incontinence episodes/24 hrs | 52 weeks
Changes from baseline in the mean number of urge incontinence episodes/24 hrs | 52 weeks
Changes from baseline in the mean number of nocturnal urinations | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Chair — Astellas Pharma Inc
Locations (2):
- Japan (2):
  - Kansai
  - Kantou

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Link to results on Astellas Clinical Study Results Web site — https://www.astellasclinicalstudyresults.com/hcp/study.aspx?ID=178-CL-051